CLINICAL TRIAL: NCT01130974
Title: A Study to Assess the Safety and Efficacy of a Daily Disposable Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 639
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bausch & Lomb contact lens (Experimental): Bausch & Lomb daily disposable cosmetic tint contact lens
  Interventions: Device: Bausch & Lomb contact lens
- Marketed daily disposable contact lens (Active Comparator): Marketed daily disposable cosmetic tint contact lens
  Interventions: Device: Marketed daily disposable contact lens

INTERVENTIONS:
Device: Bausch & Lomb contact lens — Bausch & Lomb daily disposable cosmetic tint contact lens
  Arms: Bausch & Lomb contact lens
Device: Marketed daily disposable contact lens — Marketed daily disposable cosmetic tint contact lens
  Arms: Marketed daily disposable contact lens

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the Bausch & Lomb daily disposable tint contact lens (Test) compared to a currently marketed daily disposable cosmetic tint contact lens (Control).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be adapted wearers of soft contact lenses, wear a lens in each eye, and each lens must be of the same manufacture and brand.
* Subjects must be correctable through spherocylindrical refraction to 32 letters (0.3 logMAR) or better (distance, high contrast) in each eye.
* Subjects must be of Asian descent.
* Subjects must require plano or myopic correction and must require contact lens correction from plano to -6.00 D in both eyes.

Exclusion Criteria:

* Subjects who have any systemic disease affecting ocular health.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects with an active ocular disease or are using any ocular medication.
* Subjects with any "Present" finding during the slit lamp examination that, in the Investigator's judgment, interferes with contact lens wear.
* Subjects with any scar or neovascularization within the central 4 mm of the cornea. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment, does not interfere with contact lens wear, are eligible for this study.
* Subjects who currently wear monovision, multifocal, or toric contact lenses.
* Subjects who are adapted wearers of 1-Day Acuvue Define daily disposable cosmetic tint contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bev Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 Asian participants (400 eyes) who were adapted wearers of soft contact lenses were enrolled in this 1-month study at approximately 10 investigative sites in Asia and the United States. First participant was enrolled 4/12/2010 and last participant exited the study 08/09/2010
Pre-assignment Details: Of the 200 participants (400 eyes) enrolled and dispensed lenses, 172 participants (344 eyes) completed the study
Period: Overall Study
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Started | 100 | 100
Completed | 85 | 87
Not Completed | 15 | 13
Not completed — Protocol Violation | 10 | 10
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligibility criteria | 5 | 2

BASELINE CHARACTERISTICS:
Population: All participants were randomized and dispensed lenses at the baseline visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Customized [Number; unit: participants]
  Between 18 and 62 years | 100 | 100 | 200
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 76 | 150
  Male | 26 | 24 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  Asian Decent | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings
Description: Graded Slit lamp findings (epithelial edema, epithelial microcysts, corneal staining, limbal injection, bulbar injection, upper lid tarsal conjunctival abnormalities, corneal neovascularization, and corneal infiltrates) > grade 2 over all follow-up visits, summarizes the worst case over all follow-up visits. Graded 0-4 with 0=none and 4=severe
Time Frame: Summarized over all follow-up visits through 1 month
Population: All dispensed eyes with any slit lamp findings > grade 2
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Number analyzed (Participants) | 99 | 99
Number analyzed (eyes) | 198 | 198
eyes | 0 | 0

2. Primary Outcome: logMAR Visual Acuity (VA)
Description: Non-inferiority of distance high contrast logMAR lens VA. A negative value indicates improved VA. Lens VA was established for All Study, Dispensed, 2-Week Follow-up Visit, and 1-Month Follow-up Visit
Time Frame: Summarized over all visits, and dispensed visit
Population: All eligible, dispensed eyes
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Number analyzed (Participants) | 86 | 88
Number analyzed (eyes) | 172 | 176
logMAR
  All study visits | 0.006 (0.039) | -0.009 (0.039)
  Dispensed visit | 0.006 (0.048) | -0.010 (0.048)

3. Secondary Outcome: Lens Wettability
Description: Lens wettability was rated as Grade 4-0. Grade 4 = 100% of anterior surface wettable (optimal); Grade 3 = presence of small (< 0.1 mm), individual, discrete non-wetting areas (slight); Grade 2 = presence of single area of non-wetting between 0.1 mm and 0.5 mm in size (mild); Grade 1 = presence of several areas on non-wetting, each between 0.1 mm and 0.5 mm in size (moderate); Grade 0 = presence of one or more non-wetting areas > 0.5 mm in size (severe). Suboptimal lens wettability was defined as a rating other than Grade 4, ie slight, mild, moderate, or severe ratings. Over All Visits summarizes the worst case over the dispensing and all follow-up visits.
Time Frame: Summarized over all follow-up visits through 1 month
Population: All Eligible, Dispensed Eyes, Over All Visits summarizes the worst case over the dispensing and all follow-up visits.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Marketed Contact Lens: Marketed daily disposable cosmetic tint contact lens
Arm/Group | Bausch & Lomb Contact Lens | Marketed Contact Lens
Number analyzed (Participants) | 86 | 88
Number analyzed (eyes) | 172 | 176
eyes
  Optimal | 129 | 134
  Slight | 41 | 39
  Mild | 2 | 3
  Moderate | 0 | 0
  Severe | 0 | 0

4. Secondary Outcome: Lens Deposits
Description: Degree of lens deposits was assessed as none, light, medium, or heavy. Suboptimal lens deposits were defined as a degree rating of medium or heavy. Measured over all visits through one month
Time Frame: Summarized over all follow-up visits through one month
Population: All Eligible, Dispensed Eyes, Over All Visits summarizes the worst case over the dispensing and all follow-up visits.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Contact Lens
Number analyzed (Participants) | 86 | 87
Number analyzed (eyes) | 172 | 174
eyes
  None | 152 | 151
  Light | 20 | 23
  Medium | 0 | 0
  Heavy | 0 | 0

5. Secondary Outcome: Lens Centration
Description: Lens centration was assessed as excellent(fully centered), good (slight decentration, no corneal exposure), fair (decentration, intermittent corneal exposure), or poor (incomplete corneal coverage and/or edge lift).
  Suboptimal lens centration was defined as a rating other than excellent.
Time Frame: Summarized over all follow-up visits through 1 month
Population: All Eligible, Dispensed Eyes, Over All Visits summarizes the worst case over the dispensing and all follow-up visits.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Contact Lens
Number analyzed (Participants) | 86 | 88
Number analyzed (eyes) | 172 | 176
eyes
  Excellent | 127 | 129
  Good | 31 | 26
  Fair | 13 | 6
  Poor | 1 | 15

6. Secondary Outcome: Lens Movement
Description: Lens movement was assessed as adequate, excessive (> 0.6 mm), insufficient (< 0.2 mm), or adherence. Suboptimal lens movement was defined as a rating other than adequate.
Time Frame: Summarized over all follow-up visits through one month
Population: All Eligible, Dispensed Eyes, Over All Visits summarizes the worst case over the dispensing and all follow-up visits.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Contact Lens
Number analyzed (Participants) | 86 | 88
Number analyzed (eyes) | 172 | 176
eyes
  Adequate | 167 | 152
  Excessive | 0 | 18
  Insufficient | 5 | 6
  Adherence | 0 | 0

7. Secondary Outcome: Symptoms & Complaints
Description: Subject symptoms/complaints were assessed on a scale from 0 to 100, with 0 denoting least favorable symptoms/complaints and 100 being the most favorable score.
Time Frame: Summarized over all follow-up visits through one month
Population: All eligible dispensed eyes, summarized over all follow-up visits through 1 month.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Number analyzed (Participants) | 86 | 88
Number analyzed (eyes) | 172 | 176
units on a scale
  Burning Stinging Upon Insertion | 90.3 (12.9) | 84.6 (12.9)
  Comfort | 87.1 (13.1) | 83.1 (13.1)
  End of Day Comfort | 82.0 (15.1) | 77.3 (15.1)
  Lens Awareness | 88.7 (12.9) | 80.6 (12.9)
  Lens Cleanliness | 91.9 (8.4) | 89.2 (8.4)
  Irritation | 87.4 (12.9) | 82.8 (12.9)
  Itching | 89.3 (13.3) | 84.6 (13.3)
  Dryness | 82.1 (15.7) | 77.9 (15.6)
  Redness | 89.4 (12.8) | 85.4 (12.8)
  Vision | 89.6 (11.4) | 87.9 (11.4)
  Lens Handling Upon Insertion | 89.2 (13.0) | 83.3 (13.0)
  Lens Handling Upon Removal | 92.1 (10.1) | 87.9 (10.1)
  Overall Impression | 87.5 (12.8) | 80.1 (12.8)

8. Primary Outcome: logMAR Visual Acuity (VA)
Description: as for outcome 2
Time Frame: 2 week and 1 month follow-up
Population: All eligible, dispensed eyes
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Number analyzed (Participants) | 85 | 87
Number analyzed (eyes) | 170 | 174
logMAR
  2 week visit | 0.010 (0.046) | -0.004 (0.046)
  1 month visit | 0.003 (0.043) | -0.013 (0.043)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Bausch & Lomb Contact Lens | Marketed Daily Disposable Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data generated as a result of this study will be regarded as confidential, until appropriate analysis and review by the Sponsor or its designee are completed. The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor,and such that confidential or proprietary information is not disclosed.